CLINICAL TRIAL: NCT02707302
Title: Iodophor-impregnated Versus Iodophor-free Adhesive Drapes for Prevention and Healing of Wound Infections After Total Hip Arthroplasty
Brief Title: Surgical Adhesive Drapes for Prevention and Healing of Wound Infections After Total Hip Arthroplasty
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Third Affiliated Hospital of Guangzhou University of Traditional Chinese Medicine (Industry)
Responsible Party: Principal Investigator, Zhuo Wu, Director, Third Affiliated Hospital of Guangzhou University of Traditional Chinese Medicine
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: gztcm_001
Record Dates: First submitted 2016-03-02; First posted 2016-03-14 (Estimated); Last update posted 2016-03-14 (Estimated); Status verified 2016-03

CONDITIONS: Hip Replacement

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Iodophor-impregnated adhesive drapes (Experimental): In the iodophor-impregnated adhesive drapes group, routine disinfection will be carried out and bacteria samples will be harvested 1 cm from the wound site using sterilized swabs prior to use of the surgical adhesive drapes, and again at the end of surgery before skin suturing, for preoperative bacterial culture. The packaging of the 3M™ iodophor-impregnated adhesive drapes will be opened and the aseptic adhesive drapes unfolded until the "stop" instruction. The adhesive drapes will then be pasted to the surgical wound and smoothed using an aseptic cloth, taking care to avoid air bubbles.
  Interventions: Device: Iodophor-impregnated adhesive drapes group
- Iodophor-free adhesive drapes (Experimental): Patients in the iodophor-free adhesive drapes group will undergo the same procedures, but with iodophor-free drapes.
  Interventions: Procedure: Iodophor-free adhesive drapes group

INTERVENTIONS:
Device: Iodophor-impregnated adhesive drapes group — Odd-numbered patients are randomized to the iodophor-impregnated adhesive drapes group.3M™ loban™2 iodophor-impregnated adhesive drape(3M Company, St. Paul, Minnesota, USA) will be used at the surgical site in the iodophor-impregnated adhesive drapes group.
  Arms: Iodophor-impregnated adhesive drapes
Procedure: Iodophor-free adhesive drapes group — Even-numbered patients are randomized to the iodophor-free adhesive drapes group. Iodophor-free aseptic adhesive drapes(3M Company, St. Paul, Minnesota, USA) will be used at the surgical site in the iodophor-free adhesive drapes group.
  Arms: Iodophor-free adhesive drapes

SUMMARY:
The purpose of this study is to support the rational use of iodophor-impregnated surgical adhesive drapes for preventing wound infections after total hip arthroplasty.

DETAILED DESCRIPTION:
Surgical-site infections, including deep-layer and superficial-layer wound infections, are common complications after total hip arthroplasty. Surgical infections lead to poor wound healing, increased hospital days, increased patient suffering and distress, higher costs, and even life-threatening events. Wound infections after total hip arthroplasty result in local pain, joint displacement, and reduced joint function. Compared with common bacterial infections, bacteria in the deep layer of the epidermis after total hip arthroplasty adhere to the metal prosthesis and bone cement, and may thus escape the immune system because of a lack of blood supply. Furthermore, the immune response contributes to the formation of a protective mucus layer on the prosthesis surface, and bacteria in this mucus layer may be protected from antibiotic intervention. Preventing surgical-site infection is thus an important factor determining the success of total hip arthroplasty. Measures to prevent surgical-site infection currently include instrument sterilization, protection of an aseptic area, and use of prophylactic antibacterial drugs, while reduced surgical-wound size and use of iodophor-impregnated antibacterial adhesive drapes have also been proposed to reduce infection.

Surgical adhesive drapes can create an aseptic area around the wound, thus reducing the bacterial content and infection incidence. Compared with conventional iodophor-free polyethylene adhesive drapes, iodophor-impregnated polyester surgical adhesive drapes are more breathable and scalable, show better compliance, and provide better skin adhesion. Iodophor-impregnated adhesive drapes attached to the sterilized surgical site can effectively inhibit intraoperative movement of bacteria, providing a persistent and effective protection against wound infection after total hip arthroplasty.

Total hip arthroplasty involves a long operation and has a high risk of wound infection. Iodophor-impregnated adhesive drapes are recommended because the iodophor-impregnated viscose persistently releases iodine ions to help maintain aseptic skin throughout surgery. Iodophor-impregnated adhesive drapes have been shown to decrease the incidence of wound infection and show broad-spectrum antibacterial activity for several hours, unaffected by body fluids and blood, compared with iodophor-free adhesive drapes. Iodophor-impregnated adhesive drapes have been reported to reduce surgical-site infection in orthopedic surgery. However, few studies have reported on the use of antibacterial surgical adhesive drapes in China, though Ling et al. reported that they decreased the incidence of surgical-site infection. However, despite evidence suggesting that 3M iodophor-impregnated antibacterial adhesive drapes can reduce bacteria at the surgical site, prevent wound infection, and promote wound healing.

Although the effects of surgical adhesive drapes on wound infection have been extensively studied, to the best of our knowledge, no clinical study has compared the effects of iodophor-impregnated and iodophor-free antibacterial adhesive drapes on wound infection caused by bacteria in the deep layer of the epidermis. We hypothesized that 3M iodophor-impregnated adhesive drapes would inhibit bacteria around the surgical wound and in the deep layer of the epidermis after total hip arthroplasty, and promote wound healing more effectively than 3M iodophor-free adhesive drapes. We aim to validate this hypothesis in a single-center, randomized, double-blinded, and controlled clinical trial.

Data collection, preservation, and monitoring Data will be collected on paper case-report forms and summarized in a table. The written records will be transferred to an electronic format using a double-data entry strategy. The trial process will be monitored by professional clinical research associates will full access to all essential documents to ensure patient safety and complete clinical data, including compliance with the informed-consent procedure, and evaluation of primary endpoints and compliance. In addition to regular site visits, the clinical research associates will also communicate with the trial center via e-mail and phone. If any patient(s) withdraws from the trial, an intention-to-treat analysis of related records should be performed, otherwise the patient's records will be deleted. The reasons for patient withdrawal should be recorded in the medical records.

Statistical analysis All data will be analyzed statistically using Statistical Product and Service Solutions 10.0 software. Quantitative baseline data will be compared using two-sample t-tests and Mann-Whitney U tests, and qualitative data using χ2 or Fisher's exact probability tests. Differences in VAS and Harris scores between the iodophor-impregnated and iodophor-free adhesive drapes groups will be evaluated by two-sample t-tests. Non-normally distributed data will be converted or comparisons of primary and secondary outcomes prior to and after interventions will be compared between the groups using two-sample t-tests. Bacterial detection rates in peri-wound tissue and grade I wound-healing rates between the two groups will be compared by χ2 tests. A level of P < 0.05 will be considered statistically significant.

ELIGIBILITY:
Inclusion Criteria:

* age ≥18 years;
* either sex;
* able to tolerate anesthesia and surgery;
* hip-joint disease causing chronic discomfort and obvious joint-function disorders (including primary or secondary coxarthrosis, avascular necrosis of the femoral head, rheumatoid arthritis involving the hip joint, ankylosing spondylitis involving the hip joint, hip fracture (in older), tumor in the bone joint, and hemophilic arthritis);
* informed consent signed by patients, relatives or guardians and approved by the Hospital Ethics Committee.

Exclusion Criteria:

* allergy to antiseptics, such as iodophor;
* scheduled surgical area with red swelling and ulceration; positive bacterial cultures in the first detection;
* participation in other clinical trials within 30 days prior to recruitment; pregnancy;
* human immunodeficiency virus type I and/or hepatitis virus infection; neurogenic disease, any disease presenting with rapid bone destruction, poor muscular strength around the hip joint, or complicated by other organ diseases; systemic or local severe bacterial infection; poor surgical tolerance;
* emotional disturbance;
* inability to complete the clinical trial because of poor compliance;
* unsuitability for the clinical trial according to the researchers.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Actual)
Dates: Start 2009-01; Primary Completion 2009-06 (Actual); Study Completion 2012-01 (Actual)

PRIMARY OUTCOMES:
bacterial detection rate in the peri-wound tissue | 48 hours
  Time to bacterial culture

SECONDARY OUTCOMES:
wound-healing time | 30 days after surgery
wound-healing grade | 30 days after surgery
  Wound-healing grade I = excellent wound healing without adverse reactions; grade II = inflammation including red swelling, sclerosis, hematoma and hydrops of the skin, but no suppuration; and grade III = wound suppuration and need for wound incision and drainage.
pain evaluated by the Visual Analog Scale (VAS) | 6 months after surgery
hip-joint function, evaluated by Harris hip score | 6 months after surgery

CONTACTS AND LOCATIONS:
Overall Officials: Zhuo Wu, Master, Principal Investigator — Hospital of Bone Injury, Guangzhou University of Traditional Chinese Medicine

IPD SHARING:
Plan to Share IPD: Undecided